CLINICAL TRIAL: NCT06945640
Title: Evaluation of the Efficacy, Safety, and Stability of the Surgical Navigation System 'RUS NE' in Robot-Assisted Partial Nephrectomy: A Retrospective and Prospective Comparative Study
Brief Title: Evaluation of 'RUS NE' in Robot-Assisted Partial Nephrectomy: Efficacy, Safety, and Stability
Acronym: HTK_002
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hutom Corp (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0278; A20250116 (Other Grant/Funding Number: Global innovative medical technology verification support at AMC)
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-04

CONDITIONS: Kidney Neoplasm; Nephrectomy; Surgical Navigation Systems; Renal Mass; Robot-assisted Urological Surgery
Keywords: Kidney Neoplasms; Nephrectomy; Image-Guided Surgery; Surgical Navigation Systems; Robot-assisted partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUS NE Group (Experimental): Individuals undergo robot-assisted partial nephrectomy using RUS NE
  Interventions: Device: RUS NE
- Standard Surgery Group (No Intervention): Individuals undergo robot-assisted partial nephrectomy without using RUS NE. The individuals of this group were selected from the historical group.

INTERVENTIONS:
Device: RUS NE — RUS NE is a surgical navigation system designed for use in robot-assisted partial nephrectomy. It reconstructs CT images into 3D models, providing visualization of tumor and vascular structures to enhance surgical precision and optimize resection planning. This system aids in reducing resection volume and improving operative outcomes by integrating anatomical insights into the surgical workflow.
  Arms: RUS NE Group

SUMMARY:
This study is a retrospective and prospective comparative study evaluating the efficacy, safety, and stability of the surgical navigation system 'RUS NE' in robot-assisted partial nephrectomy. The study aims to compare intraoperative and postoperative clinical indicators between the experimental group and the control group to verify the clinical effectiveness and stability of RUS NE. This research is conducted as part of the 2025 Corporate Verification Support Project of the Global Innovative Medical Technology Verification Support Center at Asan Medical Center (ARIS Project Number: A20250116) and is supported by the Korea Health Industry Development Institute's healthcare technology research and development program.

DETAILED DESCRIPTION:
1. Study Objectives

1. Efficacy Evaluation: Comparison of resection volume, operative time, and blood loss between the experimental group (RUS NE-assisted) and the control group (standard procedure).

   o Analysis of whether RUS NE facilitates accurate tumor localization to minimize resection margins.
2. Stability Evaluation: Validation of CT turn-around time, accuracy of 3D image reconstruction, and system functionality.

   - Assessment of the device's reliability and stability in a real surgical environment.
3. Study Methods

   * Study Design: Retrospective and prospective, single-center, comparative study.
   * Study Population: Patients scheduled for robot-assisted partial nephrectomy.
   * Study Period: From IRB approval to December 31, 2025.

     * Sample Size: 80 patients (20 in the experimental group, 60 in the control group).
     * Control group selection: Propensity Score Matching (1:3) applied to match previously treated patients.
4. Study Endpoints Primary Endpoint: Resection volume: To assess renal function preservation. Secondary Endpoints: Operative time, stage-specific time, blood loss, hospital stay, and postoperative complications.

Stability Evaluation: CT turn-around time, accuracy of 3D modeling, and adequacy of vascular and tumor reconstruction.

ELIGIBILITY:
Inclusion Criteria

[Experimental Group]

1. Patients diagnosed with renal cancer scheduled for robot-assisted partial nephrectomy using the RUS system, aged between 20 and 80 years.
2. Patients who voluntarily consent to participate in this clinical trial and sign the written informed consent form.
3. Patients with a renal tumor measuring ≤10 cm in maximum diameter on preoperative CT imaging.
4. Patients with a RENAL Nephrometry Score between 4 and 12.

[Control Group]

1. Patients diagnosed with renal cancer who underwent robot-assisted partial nephrectomy using the standard surgical method at the institution between January 1, 2020, and January 23, 2025.
2. Patients aged between 19 and 79 years.
3. Patients with a renal tumor measuring ≤10 cm in maximum diameter on preoperative CT imaging.
4. Patients with a RENAL Nephrometry Score between 4 and 12.

Exclusion Criteria [Experimental Group]

1. Patients who do not consent to participate in the clinical trial.
2. Patients whose CT examination does not follow the required protocol for image analysis.
3. Patients with a history of abdominal surgery likely to cause severe adhesions.
4. Patients with a solitary kidney or horseshoe kidney as identified on preoperative CT.
5. Patients scheduled for bilateral nephrectomy.
6. Patients requiring simultaneous resection of other organs in addition to nephrectomy.
7. Patients with a history of abdominal surgery where severe adhesions are expected based on the investigator's judgment.
8. Patients with severe renal dysfunction at the time of screening (serum creatinine level ≥1.5 times the upper limit of normal for the study site) or CKD stage 3 (eGFR <60).
9. Patients classified as ASA (American Society of Anesthesiologists Physical Status Classification) IV-VI.
10. Patients with a history of psychiatric disorders, alcohol abuse, or other conditions that, in the investigator's judgment, make clinical trial participation inappropriate.
11. Patients who have participated in or are scheduled to participate in another clinical trial (medical device or pharmaceutical) within four weeks prior to screening.
12. Patients deemed unsuitable for clinical trial participation at the investigator's discretion.
13. Patients whose CT images are not suitable for generating 3D images for use with the investigational medical device.

[Control Group]

1. Patients whose CT data are unavailable.
2. Patients with a history of abdominal surgery with expected or confirmed severe adhesions.
3. Patients with a solitary kidney or horseshoe kidney.
4. Patients who have undergone bilateral nephrectomy.
5. Patients who have undergone simultaneous resection of other organs in addition to nephrectomy.
6. Patients with renal dysfunction (serum creatinine level ≥1.5 times the upper limit of normal for the study site) or CKD stage 3 (eGFR <60).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Resection volume | At the time of surgery
  Resection volume were measured by ellipsoid formula. The maximum longitudinal length of the resected kidney specimen is measured along the X-axis, with perpendicular measurements taken along the Y and Z axes. The volume is estimated using the formula: (π/6) × X × Y × Z.

SECONDARY OUTCOMES:
Operative time | At the time of surgery
  The total amount time for robot-assisted partial nephrectomy, including the time for surgical console manipulation

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided